CLINICAL TRIAL: NCT04498182
Title: A Phase 2b Study Evaluating the Safety and Efficacy of AR-15512 Ophthalmic Solution for the Treatment of Dry Eye Disease (COMET-1)
Brief Title: A Phase 2b Study Evaluating the Safety and Efficacy of AR-15512 Ophthalmic Solution for the Treatment of Dry Eye Disease
Acronym: COMET-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-15512-CS201
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AR-15512 Ophthalmic Solution Higher Dose (Experimental): AR-15512 Ophthalmic Solution 0.003%, one drop in each eye twice daily for 84 days. Both eyes will be treated.
  Interventions: Drug: AR-15512 Ophthalmic Solution
- AR-15512 Ophthalmic Solution Lower Dose (Experimental): AR-15512 Ophthalmic Solution 0.0014%, one drop in each eye twice daily for 84 days. Both eyes will be treated.
  Interventions: Drug: AR-15512 Ophthalmic Solution
- Vehicle (Placebo Comparator): AR-15512 Ophthalmic Solution Vehicle, one drop in each eye twice daily for 84 days. Both eyes will be treated.
  Interventions: Drug: AR-15512 Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: AR-15512 Ophthalmic Solution — Ophthalmic solution administered via topical ocular instillation in one of two dose concentrations: 0.0014% (lower dose) or 0.003% (higher dose)
  Arms: AR-15512 Ophthalmic Solution Higher Dose; AR-15512 Ophthalmic Solution Lower Dose
Drug: AR-15512 Ophthalmic Solution Vehicle — Ophthalmic solution vehicle administered via topical ocular instillation
  Arms: Vehicle

SUMMARY:
This is a Phase 2b, multicenter, vehicle-controlled, double-masked, randomized study. All subjects enrolled will have dry eye disease. The study consists of Screening and Baseline visits to determine eligibility, followed by efficacy assessments at Day 14 (Visit 3), 28 (Visit 4) and 84 (Visit 5/Study Exit). Safety will be assessed at all study visits.

DETAILED DESCRIPTION:
At the end of the Screening Visit, all qualified subjects will be assigned to administer AR-15512 vehicle twice a day to both eyes for 14 days (vehicle run-in period). After the vehicle run-in period, subjects will be re-evaluated for signs and symptoms of Dry Eye Disease (DED). Subjects who requalify based on inclusion/exclusion criteria will be randomized in a 1:1:1 ratio to receive AR-15512 0.0014% (lower dose), AR-15512 0.003% (higher dose) or AR-15512 vehicle administered as 1 drop in each eye twice daily for 84 days.

This study will utilize a Controlled Adverse Environment (CAE) chamber, which serves to (1) minimize the factors that could impact the evaluation (temperature, humidity, and airflow) and (2) stress the ocular surface in a safe, standardized, controlled, and reproducible manner. Subjects will be exposed to the CAE for approximately 90 minutes during each CAE visit. Subjects will be exposed to the CAE at the Screening and Baseline visits as well as on Day 28 (Visit 4) and Day 84 (Visit 5). Efficacy endpoints will be evaluated pre- and post- exposure to the CAE.

Aerie Pharmaceuticals was acquired by Alcon on November 22, 2022.

ELIGIBILITY:
Key Inclusion Criteria:

* Previous history of dry eye disease (DED) within the previous 6 months;
* Have used and/or desired to use artificial tears for DED symptoms within 2 months prior to the Screening visit;
* Signs and symptoms of DED at the Screening and Baseline visits;
* Best Corrected Visual Acuity (BCVA) of 20/200 (+0.70 LogMAR) or better in both eyes at both the Screening and Baseline visits;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* History or presence of any ocular disorder or condition (other than DED) in either eye that would, in the opinion of the investigator, likely interfere with the interpretation of the study results or subject safety;
* Current evidence of other significant ophthalmic diseases which, in the opinion of the investigator, may interfere with study findings or interpretation;
* Use of contact lenses in either eye within 7 days prior to the Screening visit or planned use during the study;
* Regular use of ocular medications or nutritional supplements as specified in the protocol within 30 days prior to the Screening visit;
* Positive pregnancy test at Screening or Baseline visits or currently breastfeeding.
* Other protocol-specified exclusion criteria may apply.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scientific Advisor, Clinical Research and Development, Study Director — Alcon Research, LLC
Locations (15):
- United States (15):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Eye Research Foundation, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Midwest Cornea Associates, LLC, Carmel, Indiana
  - Michael Washburn Center for Ophthalmic Research, LLC, Indianapolis, Indiana
  - The Eye Care Institute, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - Andover Eye Associates, Raynham, Massachusetts
  - Complete Eye Care of Medina, Hamel, Minnesota
  - Moyes Eye Center, Kansas City, Missouri
  - Vita Eye Clinic, Shelby, North Carolina
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, LLC, Smyrna, Tennessee
  - Alpine Research Organization, Inc,, Clinton, Utah
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 15 clinical sites located in the United States.
Pre-assignment Details: This reporting group includes all randomized participants.
Units Other Than Participants: eyes
Groups:
- AR-15512 Ophthalmic Solution Higher Dose: AR-15512 Ophthalmic Solution 0.003%, one drop in each eye twice daily for 84 days. Both eyes were treated.
- AR-15512 Ophthalmic Solution Lower Dose: AR-15512 Ophthalmic Solution 0.0014%, one drop in each eye twice daily for 84 days. Both eyes were treated.
- Vehicle: AR-15512 Ophthalmic Solution Vehicle, one drop in each eye twice daily for 84 days. Both eyes were treated.
Period: Overall Study
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Started | 122; 244 eyes | 121; 242 eyes | 126; 252 eyes
Completed | 115; 230 eyes | 114; 228 eyes | 116; 232 eyes
Not Completed | 7; 14 eyes | 7; 14 eyes | 10; 20 eyes
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Withdrawal of Consent | 3 | 4 | 3
Not completed — Non-Compliant | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Investigator Decision | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle | Total
Number analyzed (Participants) | 122 | 121 | 126 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.01) | 65.5 (10.89) | 63.1 (11.90) | 63.7 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 82 | 92 | 266
  Male | 30 | 39 | 34 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10 | 20
  Not Hispanic or Latino | 116 | 117 | 116 | 349
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaska Native | 0 | 0 | 2 | 2
  Asian | 11 | 8 | 7 | 26
  Black / African American | 18 | 15 | 18 | 51
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 92 | 97 | 99 | 288
  Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in Pre-CAE (Controlled Adverse Environment) Ocular Discomfort Score (ODS) on a Visual Analogue Scale at Day 28
Description: Ocular discomfort was assessed using a Visual Analogue Scale (VAS) that ranged from 0 millimeters (mm) (no ocular discomfort) to 100 mm (maximum ocular discomfort). Ocular discomfort was assessed at Baseline prior to CAE exposure and at Day 28 prior to CAE exposure. The Day 28 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes. This is a co-primary endpoint.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: Intent-to-Treat (ITT) with data at both visits
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 118 | 119 | 119
millimeter (mm) | -15.3 (2.14) | -11.0 (2.12) | -11.9 (2.15)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.2305, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.4, 95% CI 2-sided [-8.9 to 2.2], Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.7436, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.9, 95% CI 2-sided [-4.6 to 6.4], Standard Error of Mean 2.81

2. Primary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Anesthetized Schirmer Test Score at Day 28
Description: The Schirmer test measures tear production. Following instillation of topical anesthetic drops, Schirmer strips were placed on the lower eye lids, eyes were closed, and strips remained in place for 5 minutes or until both strips reached a maximum score. The strips were removed, and the amount of wetting was recorded on a scale from 0 mm (no tear production) to 35 mm (maximum tear production). The test was performed at Baseline prior to CAE exposure and at Day 28 prior to CAE exposure. The Day 28 value was subtracted from the Baseline value. A more positive change value indicates a better outcome. One eye (study eye) contributed data to the analysis. This is a co-primary endpoint.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 117 | 116 | 118
Number analyzed (eyes) | 117 | 116 | 118
mm | 2.2 (0.53) | 3.0 (0.53) | 2.7 (0.53)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.4936, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.5, 95% CI 2-sided [-1.9 to 0.9], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.7131, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.3, 95% CI 2-sided [-1.1 to 1.6], Standard Error of Mean 0.70

3. Secondary Outcome: Least Squares Mean Pre-CAE Ocular Discomfort Score (ODS) on a Visual Analogue Scale at Day 28
Description: Ocular discomfort was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular discomfort) to 100 mm (maximum ocular discomfort) prior to CAE exposure. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Day 28
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 118 | 119 | 119
mm | 57.8 (2.14) | 62.1 (2.12) | 61.2 (2.15)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.2305, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.4, 95% CI 2-sided [-8.9 to 2.2], Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.7436, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.9, 95% CI 2-sided [-4.6 to 6.4], Standard Error of Mean 2.81

4. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Ocular Discomfort Score (ODS) on a Visual Analogue Scale at Day 84
Description: Ocular discomfort was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular discomfort) to 100 mm (maximum ocular discomfort). Ocular discomfort was assessed at Baseline prior to CAE exposure and at Day 84 prior to CAE exposure. The Day 84 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
mm | -20.6 (2.40) | -13.3 (2.40) | -13.6 (2.42)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0281, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -7.0, 95% CI 2-sided [-13.2 to -0.8], Standard Error of Mean 3.17
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9186, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.3, 95% CI 2-sided [-5.9 to 6.6], Standard Error of Mean 3.18

5. Secondary Outcome: Least Squares Mean Pre-CAE Ocular Discomfort Score (ODS) on a Visual Analogue Scale at Day 84
Description: as for outcome 3
Time Frame: Day 84
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
mm | 52.4 (2.40) | 59.7 (2.40) | 59.4 (2.42)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0281, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -7.0, 95% CI 2-sided [-13.2 to -0.8], Standard Error of Mean 3.17
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9186, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.3, 95% CI 2-sided [-5.9 to 6.6], Standard Error of Mean 3.18

6. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Anesthetized Schirmer Test Score at Day 84
Description: The Schirmer test measures tear production. Following instillation of topical anesthetic drops, Schirmer strips were the placed on the lower eye lids, eyes were closed, and strips remained in place for 5 minutes or until both strips reached a maximum score. The strips were removed, and the amount of wetting was recorded on a scale from 0 mm (no tear production) to 35 mm (maximum tear production). The test was performed at Baseline prior to CAE exposure and at Day 84 prior to CAE exposure. The Day 84 value was subtracted from the Baseline value. A more positive change value indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
Number analyzed (eyes) | 115 | 114 | 116
mm | 2.9 (0.57) | 3.2 (0.56) | 2.9 (0.57)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.9846, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.0, 95% CI 2-sided [-1.5 to 1.5], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.6508, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.3, 95% CI 2-sided [-1.1 to 1.8], Standard Error of Mean 0.75

7. Secondary Outcome: Least Squares Mean Pre-CAE Anesthetized Schirmer Test Score at Day 84
Description: The Schirmer test measures tear production. Following instillation of topical anesthetic drops, Schirmer strips were the placed on the lower eye lids, eyes were closed, and strips remained in place for 5 minutes or until both strips reached a maximum score. The strips were removed, and the amount of wetting was recorded on a scale from 0 mm (no tear production) to 35 mm (maximum tear production). A higher score indicates a better outcome. The test was performed prior to CAE exposure. One eye (study eye) contributed data to the analysis.
Time Frame: Day 84
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
Number analyzed (eyes) | 115 | 114 | 116
mm | 7.9 (0.57) | 8.2 (0.56) | 7.9 (0.57)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.9846, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.0, 95% CI 2-sided [-1.5 to 1.5], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.6508, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.3, 95% CI 2-sided [-1.1 to 1.8], Standard Error of Mean 0.75

8. Secondary Outcome: Least Squares Mean Pre-CAE Anesthetized Schirmer Test Score at Day 28
Description: as for outcome 7
Time Frame: Day 28
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 117 | 116 | 118
Number analyzed (eyes) | 117 | 116 | 118
mm | 7.2 (0.53) | 7.9 (0.53) | 7.7 (0.53)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.4936, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.5, 95% CI 2-sided [-1.9 to 0.9], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.7131, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.3, 95% CI 2-sided [-1.1 to 1.6], Standard Error of Mean 0.70

9. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Pain Score on a Visual Analogue Scale at Day 84
Description: Ocular pain was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain). Ocular pain was assessed at Baseline prior to CAE exposure and at Day 84 prior to CAE exposure. The Day 84 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
mm | -18.3 (2.55) | -12.6 (2.57) | -12.4 (2.58)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0786, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -6.0, 95% CI 2-sided [-12.6 to 0.7], Standard Error of Mean 3.38
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9477, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.2, 95% CI 2-sided [-6.9 to 6.5], Standard Error of Mean 3.39

10. Secondary Outcome: Least Squares Mean Pre-CAE Pain Score on a Visual Analogue Scale at Day 84
Description: Ocular pain was assessed prior to CAE exposure using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain) prior to CAE exposure. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Day 84
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
mm | 36.1 (2.55) | 41.8 (2.57) | 42.1 (2.58)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0786, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -6.0, 95% CI 2-sided [-12.6 to 0.7], Standard Error of Mean 3.38
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9477, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.2, 95% CI 2-sided [-6.9 to 6.5], Standard Error of Mean 3.39

11. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Pain Score on a Visual Analogue Scale at Day 28
Description: Ocular pain was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain). Ocular pain was assessed at Baseline prior to CAE exposure and at Day 28 prior to CAE exposure. The Day 28 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 118 | 119 | 119
mm | -11.6 (2.39) | -6.6 (2.39) | -6.6 (2.41)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.1153, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Means Difference = -5.0, 95% CI 2-sided [-11.2 to 1.2], Standard Error of Mean 3.16
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9975, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.0, 95% CI 2-sided [-6.2 to 6.2], Standard Error of Mean 3.15

12. Secondary Outcome: Least Squares Mean Pre-CAE Pain Score on a Visual Analogue Scale at Day 28
Description: as for outcome 10
Time Frame: Day 28
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 118 | 119 | 119
mm | 43.0 (2.39) | 48.0 (2.39) | 48.0 (2.41)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.1153, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -5.0, 95% CI 2-sided [-11.2 to 1.2], Standard Error of Mean 3.16
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9975, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.0, 95% CI 2-sided [-6.2 to 6.2], Standard Error of Mean 3.15

13. Secondary Outcome: Least Squares Mean Change From Baseline in Post-CAE Pain Score on a Visual Analogue Scale at Day 84
Description: Ocular pain was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain). Ocular pain was assessed at Baseline prior to CAE exposure and at Day 84 following CAE exposure. The Day 84 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 103 | 97 | 94
mm | -17.6 (2.77) | -8.9 (2.85) | -12.1 (2.93)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.1518, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -5.5, 95% CI 2-sided [-13.0 to 2.0], Standard Error of Mean 3.82
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.4070, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 3.2, 95% CI 2-sided [-4.4 to 10.8], Standard Error of Mean 3.87

14. Secondary Outcome: Least Squares Mean Post-CAE Pain Score on a Visual Analogue Scale at Day 84
Description: Ocular pain was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain) following CAE exposure. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Day 84
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 103 | 97 | 94
mm | 50.0 (2.77) | 58.7 (2.85) | 55.5 (2.93)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.1518, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -5.5, 95% CI 2-sided [-13.0 to 2.0], Standard Error of Mean 3.82
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.4070, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 3.2, 95% CI 2-sided [-4.4 to 10.8], Standard Error of Mean 3.87

15. Secondary Outcome: Least Squares Mean Change From Baseline in Post-CAE Pain Score on a Visual Analogue Scale at Day 28
Description: Ocular pain was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain). Ocular pain was assessed at Baseline prior to CAE exposure and at Day 28 following CAE exposure. The Day 28 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 104 | 97 | 101
mm | -7.5 (2.64) | -7.2 (2.70) | -6.4 (2.71)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.7560, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -1.1, 95% CI 2-sided [-8.1 to 5.9], Standard Error of Mean 3.56
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.8308, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.8, 95% CI 2-sided [-7.9 to 6.4], Standard Error of Mean 3.62

16. Secondary Outcome: Least Squares Mean Post-CAE Pain Score on a Visual Analogue Scale at Day 28
Description: as for outcome 14
Time Frame: Day 28
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 104 | 97 | 101
mm | 59.7 (2.64) | 60.0 (2.70) | 60.8 (2.71)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.7560, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -1.1, 95% CI 2-sided [-8.1 to 5.9], Standard Error of Mean 3.56
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.8308, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.8, 95% CI 2-sided [-7.9 to 6.4], Standard Error of Mean 3.62

17. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Global SANDE Questionnaire Score at Day 28
Description: The SANDE questionnaire assesses the frequency and severity of dry eye disease symptoms. Subjects used 2 unique, 100 mm Visual Analogue Scales (VAS) to mark the frequency of symptoms (0=rarely, 100=all the time) and the severity of symptoms (0=very mild, 100=very severe) for both eyes together. The Global SANDE score was calculated by multiplying the frequency score by the severity score and obtaining the square root. The final value was rounded nearest whole number. The SANDE questionnaire was completed at Baseline prior to CAE exposure and at Day 28 prior to CAE exposure. The Day 28 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 118 | 119 | 117
mm | -12.9 (1.70) | -9.3 (1.69) | -5.0 (1.72)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0005, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -7.9, 95% CI 2-sided [-12.4 to -3.5], Standard Error of Mean 2.26
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.0585, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -4.3, 95% CI 2-sided [-8.7 to 0.2], Standard Error of Mean 2.26

18. Secondary Outcome: Least Squares Mean Pre-CAE Global SANDE Questionnaire Score at Day 28
Description: The SANDE questionnaire assesses the frequency and severity of dry eye disease symptoms. Subjects used 2 unique, 100 mm Visual Analogue Scales (VAS) to mark the frequency of symptoms (0=rarely, 100=all the time) and the severity of symptoms (0=very mild, 100=very severe) for both eyes together. The Global SANDE score was calculated by multiplying the frequency score by the severity score and obtaining the square root. The final value was rounded nearest whole number. The SANDE questionnaire was completed prior to CAE exposure. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Day 28
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 118 | 119 | 118
mm | 62.8 (1.70) | 66.5 (1.69) | 70.8 (1.72)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0005, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -7.9, 95% CI 2-sided [-12.4 to -3.5], Standard Error of Mean 2.26
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.0585, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -4.3, 95% CI 2-sided [-8.7 to 0.2], Standard Error of Mean 2.26

19. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Global SANDE Questionnaire Score at Day 84
Description: The SANDE questionnaire assesses the frequency and severity of dry eye disease symptoms. Subjects used 2 unique, 100 mm Visual Analogue Scales (VAS) to mark the frequency of symptoms (0=rarely, 100=all the time) and the severity of symptoms (0=very mild, 100=very severe) for both eyes together. The Global SANDE score was calculated by multiplying the frequency score by the severity score and obtaining the square root. The final value was rounded nearest whole number. The SANDE questionnaire was completed at Baseline prior to CAE exposure and at Day 84 prior to CAE exposure. The Day 84 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 115
mm | -17.2 (2.09) | -9.5 (2.09) | -8.3 (2.12)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0015, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -8.9, 95% CI 2-sided [-14.3 to -3.4], Standard Error of Mean 2.77
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.6812, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -1.1, 95% CI 2-sided [-6.6 to 4.3], Standard Error of Mean 2.78

20. Secondary Outcome: Least Squares Mean Pre-CAE Global SANDE Questionnaire Score at Day 84
Description: as for outcome 18
Time Frame: Day 84
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
mm | 58.6 (2.09) | 66.3 (2.09) | 67.5 (2.12)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0015, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -8.9, 95% CI 2-sided [-14.3 to -3.4], Standard Error of Mean 2.77
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.6812, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -1.1, 95% CI 2-sided [-6.6 to 4.3], Standard Error of Mean 2.78

21. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Eye Dryness Score on a Visual Analogue Scale at Day 28
Description: Eye dryness was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no eye dryness) to 100 mm (maximum eye dryness). Eye dryness was assessed at Baseline prior to CAE exposure and at Day 28 prior to CAE exposure. The Day 28 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 117 | 118 | 119
mm | -11.3 (1.91) | -8.2 (1.90) | -7.8 (1.91)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose; Test type: Superiority; p = 0.1520, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.6, 95% CI 2-sided [-8.5 to 1.3], Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.8515, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.5, 95% CI 2-sided [-5.4 to 4.4], Standard Error of Mean 2.49

22. Secondary Outcome: Least Squares Mean Pre-CAE Eye Dryness Score on a Visual Analogue Scale at Day 28
Description: Eye dryness was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no eye dryness) to 100 mm (maximum eye dryness) prior to CAE exposure. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Day 28
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 117 | 118 | 119
mm | 63.4 (1.91) | 66.5 (1.90) | 66.9 (1.91)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.1520, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.6, 95% CI 2-sided [-8.5 to 1.3], Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.8515, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.5, 95% CI 2-sided [-5.4 to 4.4], Standard Error of Mean 2.49

23. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Eye Dryness Score on a Visual Analogue Scale at Day 84
Description: Eye dryness was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no eye dryness) to 100 mm (maximum eye dryness). Eye dryness was assessed at Baseline prior to CAE exposure and at Day 84 prior to CAE exposure. The Day 84 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
mm | -17.1 (2.20) | -11.5 (2.21) | -10.8 (2.22)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0302, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -6.3, 95% CI 2-sided [-12.1 to -0.6], Standard Error of Mean 2.91
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.8013, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.7, 95% CI 2-sided [-6.5 to 5.0], Standard Error of Mean 2.92

24. Secondary Outcome: Least Squares Mean Pre-CAE Eye Dryness Score on a Visual Analogue Scale at Day 84
Description: as for outcome 22
Time Frame: Day 84
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
mm | 57.4 (2.20) | 63.0 (2.21) | 63.7 (2.22)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose; Test type: Superiority; p = 0.0302, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -6.3, 95% CI 2-sided [-12.1 to -0.6], Standard Error of Mean 2.91
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.8013, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -0.7, 95% CI 2-sided [-6.5 to 5.0], Standard Error of Mean 2.92

25. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Ocular Discomfort Score (ODS) on a Visual Analogue Scale at Day 14
Description: Ocular discomfort was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular discomfort) to 100 mm (maximum ocular discomfort). Ocular discomfort was assessed at Baseline prior to CAE exposure and at Day 14 prior to CAE exposure. The Day 14 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 14
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 124
mm | -10.1 (1.92) | -8.2 (1.92) | -10.7 (1.90)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.8166, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.6, 95% CI 2-sided [-4.4 to 5.5], Standard Error of Mean 2.52
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.3371, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 2.4, 95% CI 2-sided [-2.5 to 7.4], Standard Error of Mean 2.52

26. Secondary Outcome: Mean Change From Baseline in Pre-CAE Ora Calibra® Ocular Discomfort Score (ODS) at Day 28
Description: Ocular discomfort was assessed using a 5-point proprietary scale where 0=no discomfort and 4=constant discomfort. Ocular discomfort was assessed at Baseline prior to CAE exposure and at Day 28 prior to CAE exposure. The Day 28 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visits
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 117 | 116 | 118
Number analyzed (eyes) | 117 | 116 | 118
score on a scale | -0.4 (1.03) | -0.4 (1.02) | -0.3 (1.11)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.3365, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.7323, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Mean Change From Baseline in Pre-CAE Ora Calibra® Ocular Discomfort Score (ODS) at Day 84
Description: Ocular discomfort was assessed using a 5-point proprietary scale where 0=no discomfort and 4=constant discomfort. Ocular discomfort was assessed at Baseline prior to CAE exposure and at Day 84 prior to CAE exposure. The Day 84 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
Number analyzed (eyes) | 115 | 114 | 116
score on a scale | -0.8 (1.22) | -0.5 (1.16) | -0.5 (1.34)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.1557, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.6845, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Least Squares Mean Pre-CAE Ocular Discomfort Score (ODS) on a Visual Analogue Scale at Day 14
Description: as for outcome 3
Time Frame: Day 14
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 124
mm | 63.0 (1.92) | 64.8 (1.92) | 62.4 (1.90)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.8166, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.6, 95% CI 2-sided [-4.4 to 5.5], Standard Error of Mean 2.52
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority — Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; p = 0.3371, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 2.4, 95% CI 2-sided [-2.5 to 7.4], Standard Error of Mean 2.52

29. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Pain Score on a Visual Analogue Scale at Day 14
Description: Ocular pain was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain). Ocular pain was assessed at Baseline prior to CAE exposure and at Day 14 prior to CAE exposure. The Day 14 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 14
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 124
mm | -4.3 (2.13) | -1.8 (2.14) | -6.1 (2.11)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.5215, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 1.8, 95% CI 2-sided [-3.7 to 7.3], Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.1312, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 4.2, 95% CI 2-sided [-1.3 to 9.8], Standard Error of Mean 2.81

30. Secondary Outcome: Least Squares Mean Pre-CAE Pain Score on a Visual Analogue Scale at Day 14
Description: Ocular pain was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no ocular pain) to 100 mm (maximum ocular pain) prior to CAE exposure. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Day 14
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 124
mm | 50.3 (2.13) | 52.8 (2.14) | 48.5 (2.11)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.5215, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 1.8, 95% CI 2-sided [-3.7 to 7.3], Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.1312, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 4.2, 95% CI 2-sided [-1.3 to 9.8], Standard Error of Mean 2.81

31. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Global SANDE Questionnaire Score at Day 14
Description: The SANDE questionnaire assesses the frequency and severity of dry eye disease symptoms. Subjects used 2 unique, 100 mm Visual Analogue Scales (VAS) to mark the frequency of symptoms (0=rarely, 100=all the time) and the severity of symptoms (0=very mild, 100=very severe) for both eyes together. The Global SANDE score was calculated by multiplying the frequency score by the severity score and obtaining the square root. The final value was rounded nearest whole number. The SANDE questionnaire was completed at Baseline prior to CAE exposure and at Day 14 prior to CAE exposure. The Day 14 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 14
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 123
mm | -7.4 (1.50) | -5.9 (1.51) | -2.9 (1.50)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0254, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -4.5, 95% CI 2-sided [-8.4 to -0.6], Standard Error of Mean 1.99
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.1362, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.0, 95% CI 2-sided [-6.9 to 0.9], Standard Error of Mean 1.99

32. Secondary Outcome: Least Squares Mean Pre-CAE Global SANDE Questionnaire Score at Day 14
Description: as for outcome 18
Time Frame: Day 14
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 124
mm | 68.3 (1.50) | 69.8 (1.51) | 72.8 (1.50)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0254, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -4.5, 95% CI 2-sided [-8.4 to -0.6], Standard Error of Mean 1.99
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.1362, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.0, 95% CI 2-sided [-6.9 to 0.9], Standard Error of Mean 1.99

33. Secondary Outcome: Least Squares Mean Change From Baseline in Pre-CAE Eye Dryness Score on a Visual Analogue Scale at Day 14
Description: Eye dryness was assessed using a Visual Analogue Scale (VAS) that ranged from 0 mm (no eye dryness) to 100 mm (maximum eye dryness). Eye dryness was assessed at Baseline prior to CAE exposure and at Day 14 prior to CAE exposure. The Day 14 value was subtracted from the Baseline value. A more negative change value indicates a better outcome. This was a subject based assessment, and subject assigned a single score for both eyes.
Time Frame: Baseline (Day 1) (pre-treatment), Day 14
Population: ITT with data at both visits
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 123
mm | -8.8 (1.56) | -4.9 (1.56) | -4.9 (1.56)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0573, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.9, 95% CI 2-sided [-8.0 to 0.1], Standard Error of Mean 2.06
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9930, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.0, 95% CI 2-sided [-4.0 to 4.1], Standard Error of Mean 2.06

34. Secondary Outcome: Least Squares Mean Pre-CAE Eye Dryness Score on a Visual Analogue Scale at Day 14
Description: as for outcome 22
Time Frame: Day 14
Population: ITT with data at visit
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 120 | 120 | 123
mm | 65.7 (1.56) | 69.7 (1.56) | 69.7 (1.56)
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.0573, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = -3.9, 95% CI 2-sided [-8.0 to 0.1], Standard Error of Mean 2.06
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.9930, ANCOVA; Based on analysis of covariance (ANCOVA) models with effects of treatment, baseline, and analysis center; LS Mean Difference = 0.0, 95% CI 2-sided [-4.0 to 4.1], Standard Error of Mean 2.06

35. Secondary Outcome: Percentage of Subjects With a Baseline Anesthetized Schirmer Score Equal to or Less That 5 mm That Achieved an Anesthetized Schirmer Score of Equal to or Greater Than 10 mm at Day 84
Description: The Schirmer test measures tear production. Following instillation of topical anesthetic drops, Schirmer strips were the placed on the lower eye lids, eyes were closed, and strips remained in place for 5 minutes or until both strips reached a maximum score. The strips were removed, and the amount of wetting was recorded on a scale from 0 mm (no tear production) to 35 mm (maximum tear production). The test was performed at Baseline prior to CAE exposure and at Day 84 prior to CAE exposure. A higher percentage indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
Number analyzed (eyes) | 115 | 114 | 116
percentage of subjects | 16.5 | 13.2 | 12.1
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.3068, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.70 to 3.15]
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.6167, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.56 to 2.68]

36. Secondary Outcome: Percentage of Subjects With a Baseline Anesthetized Schirmer Score Equal to or Less That 5 mm That Achieved an Anesthetized Schirmer Score of Equal to or Greater Than 10 mm at Day 28
Description: The Schirmer test measures tear production. Following instillation of topical anesthetic drops, Schirmer strips were the placed on the lower eye lids, eyes were closed, and strips remained in place for 5 minutes or until both strips reached a maximum score. The strips were removed, and the amount of wetting was recorded on a scale from 0 mm (no tear production) to 35 mm (maximum tear production). The test was performed at Baseline prior to CAE exposure and at Day 28 prior to CAE exposure. A higher percentage indicates a better outcome. One eye (study eye) contributed data to the analysis.
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visit
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 117 | 116 | 118
Number analyzed (eyes) | 117 | 116 | 118
percentage of subjects | 10.3 | 9.5 | 13.6
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.2867, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.28 to 1.46]
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.3803, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.32 to 1.57]

37. Secondary Outcome: Percentage of Subjects That Achieved at Least a 10 mm Increase in Pre-CAE Anesthetized Schirmer Score Relative to Baseline at Day 28
Description: as for outcome 36
Time Frame: Baseline (Day 1) (pre-treatment), Day 28
Population: ITT with data at both visits
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 117 | 116 | 118
Number analyzed (eyes) | 117 | 116 | 118
percentage of subjects | 11.1 | 9.5 | 7.6
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.4375, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.58 to 3.58]
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.5840, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.51 to 3.27]

38. Secondary Outcome: Percentage of Subjects That Achieved at Least a 10 mm Increase in Pre-CAE Anesthetized Schirmer Score Relative to Baseline at Day 84
Description: as for outcome 35
Time Frame: Baseline (Day 1) (pre-treatment), Day 84
Population: ITT with data at both visits
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | AR-15512 Ophthalmic Solution Higher Dose | AR-15512 Ophthalmic Solution Lower Dose | Vehicle
Number analyzed (Participants) | 115 | 114 | 116
Number analyzed (eyes) | 115 | 114 | 116
percentage of subjects | 7.8 | 13.2 | 11.2
Statistical Analysis 1: Comparison: AR-15512 Ophthalmic Solution Higher Dose vs Vehicle; Test type: Superiority; p = 0.5046, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.29 to 1.84]
Statistical Analysis 2: Comparison: AR-15512 Ophthalmic Solution Lower Dose vs Vehicle; Test type: Superiority; p = 0.5751, Cochran-Mantel-Haenszel; Adjusted by analysis center; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.56 to 2.88]

ADVERSE EVENTS:
Time Frame: An adverse event was (AE) defined as any untoward medical occurrence associated with the administration of the drug in humans, whether or not considered drug related. AE's were collected from time of consent until study exit, approximately 14 weeks.
Description: The safety population includes all randomized subjects who have received at least one dose of the investigational product. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more arms.
Groups:
- Pretreatment: AEs reported in this group occurred prior to treatment with the study drug.
- AR-15512 Ophthalmic Solution Higher Dose - Ocular; AR-15512 Ophthalmic Solution Higher Dose - Nonocular: AEs reported in this group occurred during the AR-15512 Ophthalmic Solution 0.003% treatment period.
- AR-15512 Ophthalmic Solution Lower Dose - Ocular; AR-15512 Ophthalmic Solution Lower Dose - Nonocular: AEs reported in this group occurred during the AR-15512 Ophthalmic Solution 0.0014% treatment period.
- Vehicle - Ocular; Vehicle - Nonocular: AEs reported in this group occurred during the Vehicle treatment period.
Arm/Group | Pretreatment | AR-15512 Ophthalmic Solution Higher Dose - Ocular | AR-15512 Ophthalmic Solution Higher Dose - Nonocular | AR-15512 Ophthalmic Solution Lower Dose - Ocular | AR-15512 Ophthalmic Solution Lower Dose - Nonocular | Vehicle - Ocular | Vehicle - Nonocular
All-Cause Mortality (participants affected / at risk) | 0/369 | 0/122 | 0/122 | 0/121 | 0/121 | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/369 | 0/122 | 1/122 | 0/121 | 1/121 | 0/126 | 2/126
Other Adverse Events (participants affected / at risk) | 11/369 | 53/122 | 0/122 | 45/121 | 0/121 | 4/126 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=369) | AR-15512 Ophthalmic Solution Higher Dose - Ocular (N=122) | AR-15512 Ophthalmic Solution Higher Dose - Nonocular (N=122) | AR-15512 Ophthalmic Solution Lower Dose - Ocular (N=121) | AR-15512 Ophthalmic Solution Lower Dose - Nonocular (N=121) | Vehicle - Ocular (N=126) | Vehicle - Nonocular (N=126)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=369) | AR-15512 Ophthalmic Solution Higher Dose - Ocular (N=122) | AR-15512 Ophthalmic Solution Higher Dose - Nonocular (N=122) | AR-15512 Ophthalmic Solution Lower Dose - Ocular (N=121) | AR-15512 Ophthalmic Solution Lower Dose - Nonocular (N=121) | Vehicle - Ocular (N=126) | Vehicle - Nonocular (N=126)
Instillation site pain (General disorders) | 11 (11) | 53 (54) | 0 (0) | 45 (45) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT04498182/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT04498182/SAP_001.pdf